CLINICAL TRIAL: NCT04212182
Title: The Physiological Effect of High Flow Oxygen Therapy on Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: The Physiological Effect of High Flow Oxygen Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Rongchang Chen, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GIRH-HFNC8306
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: High-flow Nasal Cannula; Non-invasive Positive Pressure Ventilation; Acute Exacerbation of Chronic Obstructive Pulmonary Disease

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC group (Experimental): AECOPD patients receive ventilation support via HFNC.
  Interventions: Device: HFNC
- NPPV group (Active Comparator): AECOPD patients receive ventilation support via NPPV.
  Interventions: Device: NPPV

INTERVENTIONS:
Device: HFNC — HFNC provides warmed and humidified gas administered through slightly enlarged nasal prongs.
  Arms: HFNC group
Device: NPPV — NPPV is the standard therapy for ventilatory failure in AECOPD.
  Arms: NPPV group

SUMMARY:
Although non-invasive positive pressure ventilation (NPPV) shows the good curative effect of treating the patients with acute exacerbation of chronic obstructive pulmonary disease (AECOPD), some patients do not tolerate NPPV or do not benefit from it. High-flow nasal cannula (HFNC) is well tolerated and may be used to patients with AECOPD who are intolerant to NPPV treatment. This study is to evaluate the physiological effect of HFNC and compare it with NPPV.

ELIGIBILITY:
Inclusion Criteria:

* AECOPD patients with acute hypercapnic respiratory failure

Exclusion Criteria:

* other lung/pleural diseases or thoracic deformity
* severe heart failure (New York Heart Association class IV), severe dysrhythmia
* unstable angina, or malignant comorbidity
* obesity (BMI ≥ 35 kg/m²)
* severe obstructive sleep apnea syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-12-27 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Neural respiratory drive | 30 minutes
  Neural respiratory drive is calculated by diaphragm electromyogram

SECONDARY OUTCOMES:
Work of breathing | 30 minutes
  Work of breathing is calculated by the transdiaphragmatic pressure
Transcutaneous CO2 | 30 minutes
  Transcutaneous CO2 is a non-invasive method estimated the partial pressure of arterial blood CO2.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, MD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University., Guangzhou, Guangdong, China